CLINICAL TRIAL: NCT05839054
Title: Evaluation of Virtual Reality Glasses Use During Inhaler Treatment in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berker Okay, Principal Investigator, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22/197
Record Dates: First submitted 2023-04-07; First posted 2023-05-03 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Bronchiolitis; Anxiety
Keywords: Inhaler treatment; Children; Virtual reality glasses
MeSH Terms: conditions — Bronchiolitis; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The children randomize 3 different groups. A computer-generated block method divided children into 3 groups (VR glasses roller coaster, VR glasses wild dolphins, and control).
  Based on 45 randomly sorted sets (1, 2, 3) (eg Set 1 Group 2, Set 2 Group 3, Set 3 Group 1), a total of 135 unique codes were generated and then randomly placed in a blocking box. protected. Only the second researcher knew the group value of the sets.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Children were identified by a single investigator. He referred the child to the other investigator by noting the FLACC and MYPAS score, as well as the RR, SpO2, and HR values, which he determined to establish his criteria, including the first investigator. The second investigator divided the child into groups using the randomization method, with the double chronometer during the treatment, the duration of the crying and the effective treatment time were desired. He was re-directed to the first investigator, not telling the first investigator to group the treatment ending families and groups. Thus, before and after the first investigator's examination, when filling in the FLACC and MYPAS score and determining SpO2, RR and HR, the groups did not know which group they belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Roller Coasters, group 1 (Experimental): VR audio-visual users with Roller Coasters
  Interventions: Device: Virtual Reality audio and visual glass (Roller Coasters, group 1)
- Wild Dolphins, group 2 (Experimental): VR audio-visual users with Wild Dolphins
  Interventions: Device: Virtual Reality audio and visual glass (Wild Dolphins, group 2)
- group 3 (No Intervention): did not use any additional equipment

INTERVENTIONS:
Device: Virtual Reality audio and visual glass (Roller Coasters, group 1) — During the inhaler treatment, the child was shown Roller Coasters with VR glasses.
  Arms: Roller Coasters, group 1
Device: Virtual Reality audio and visual glass (Wild Dolphins, group 2) — During the inhaler treatment, the child was shown Wild Dolphins with VR glasses.
  Arms: Wild Dolphins, group 2

SUMMARY:
Virtual reality (VR) glasses are technological devices that are often used in medical fields recently and are seen as suitable for distracting children. In the last few years, many studies have been conducted to facilitate pediatric patients against painful or frightening medical procedures. For uncomfortable procedures, distracting the child's attention is seen as the most important point. VR technology has been used for procedures such as burn cases, tooth extraction, intramuscular injection, intravenous cannula, lumbar puncture, and the results of the research have been found to be satisfactory. Using VR glasses alone or in combination with standard care is effective in reducing pain and anxiety. So far, there is no study in the literature on distraction with VR during inhaler treatment in pediatric patients. Children cannot receive inhaler treatment efficiently due to reasons such as restlessness, crying, and pulling the mask during inhaler treatment, and their hospital stay is prolonged. In this study, the investigators planned to compare the patients who received inhaler treatment with VR glasses with the patients who received treatment without the aid of any device in terms of treatment compliance.

Thus, the investigators aimed to make the inhaler treatment more comfortable with VR technology.

DETAILED DESCRIPTION:
The study was designed by including children aged 2-5 years, who needed inhaler treatment (salbutamol) between 10.11.2022 and 01.04.2023, whose families gave consent for the study. This age group (preschool) was chosen because it is the age group that presents the most difficulties to families and physicians during inhaler treatment and screen exposure does not cause problems up to a certain point. The study was conducted as a prospective, single-blind, randomized, controlled study in the Pediatric Emergency Department of the Health Sciences University Haseki Training and Research Hospital.

Children with neuromotor retardation, visual and auditory problems, underlying chronic diseases (bronchiolitis, chronic lung diseases other than asthma, congenital heart diseases, neurological diseases such as epilepsy), obesity or malnutrition (to equalize the effectiveness of the drug dose), adrenaline, budesonide or Those who receive ipratropium bromide treatment, those who will receive inhaler nebula treatment for the first time, those who have received inhaler treatment in the last 72 hours, those who have a previous operation or sedative history, those who have a fever above 37.5°C, those who have used VR before, those under 2 years of age to avoid screen exposure children (infants) and children over 5 years old (school period) were excluded from the study. In addition, children with a saturation value below 92% at the time of admission, those presenting with severe asthma attacks and those with respiratory failure symptoms were not included in the study. Children with a score of 5 and above according to the bronchiolitis severity score were excluded from the study.

The children included in the study were divided into 3 groups by randomization method: VR audio-visual users (Roller Coasters, group 1), VR audio-visual users (Wild Dolphins, group 2) and those who did not use any additional equipment. (group 3). These children were observed during their 15-minute inhaler treatment and the groups were compared in terms of crying times, changes in RR, SpO2, HR values with pre- and post-treatment physician questionnaires and family questionnaires.

In the comparison study of Gerceker et al., with VR glasses in children from whom blood was drawn, the pain score was found to be 1.2 ± 2.2 in children using VR glasses, and 4.1 ± 3.5 in children without VR (control group), and the standard effect size was determined as 0.99 in the power analysis based on these data. When the number of 45 cases in each group is taken, the power of the study was calculated to be with a 1% margin of error and 98% power.

During the study period (November 2022 - April 2023), 913 children received inhaler treatment in our hospital. Children who met the selection criteria and whose families agreed to participate in the study were included in the study, and the study was terminated when the target number of 135 children was reached. 689 children who did not meet the inclusion criteria (such as chronic disease or severe bronchiolitis) and were not suitable for their age (such as under 2 years old, over 5 years old) were excluded from the study. Of the 224 children who met the inclusion criteria, 89 were excluded because they refused to participate in the study.

The children to be included in the study were determined by randomization method. For randomization, the site named randomizer.org was used to randomize 3 different groups. A computer-generated block method divided children into 3 groups (VR glasses roller coaster, VR glasses wild dolphins, and control). Based on 45 randomly sorted sets (1, 2, 3) (eg Set 1 Group 2, Set 2 Group 3, Set 3 Group 1), a total of 135 unique codes were generated and then randomly placed in a blocking box. protected. Only the second researcher knew the group value of the sets.

The children included in the study were divided into 3 groups: VR audio-visual users (Roller Coasters, group 1), VR audio-visual users (Wild Dolphins, group 2), and those who did not use any additional equipment (group 3). 3D Roller Coasters and 3D Wild Dolphins videos were used as VR images via Youtube application (Google LLC. California, USA; Youtube®). VR glasses were integrated into the tablet and given to the accompanying parent, so that the parent could see what their child was watching at that moment.

Children in all groups were given 'salbutamol' inhaler treatment for 15 minutes, and equality was achieved between the groups in terms of treatment active substance and duration. Salbutamol was given to each child as 2.5 mg/2.5 ml. The children were observed during their 15-minute inhaler treatment, and the crying times were compared with the anxiety scoring made by the same doctor before and after the treatment, and the minute respiratory rate (RR), oxygen saturation (SpO2), heart rate change (HR) and the duration of inhaler treatment were compared. In addition, families filled out questionnaires about their children's mental state before and after the treatment. The FLACC (Face, Legs, Activity, Cry, consolability) Pain Assessment Scale was used for the anxiety scoring made by the physician, and the Yale Modified Anxiety Scale (MYPAS), which was thought to be appropriate for our study, although it was designed to measure pre-operative anxiety. For families, a form consisting of eight 'yes-no' questions called the Parents' Pain Measure (MPPM), modified by us and normally used for post-operative anxiety/pain measurement, was used. In addition, Wong Baker Faces Pain Rating Scale (WBS) was also used to evaluate the anxiety of the children for convenience to the family.

The children to be included in the study were determined by a single researcher. The first investigator identified the children who met the inclusion criteria, noted the FLACC and MYPAS score, as well as the RR, SpO2, and HR values, and referred the child to the other investigator. The second investigator divided the child into his group using the randomization method, and determined the duration of crying and effective treatment, along with the duration of treatment, with a double chronometer during treatment. At the end of the treatment, the family and the child were re-directed to the first researcher on the condition that they did not tell the first researcher which group they were in. Thus, it was ensured that the first investigator did not know which group the child belonged to while filling in the FLACC and MYPAS score before and after the treatment and determining SpO2, RR and HR. In addition, with the MPPM and WBS performed by the families, the changes in the children's discomfort/restlessness were determined from the family's point of view before and after the treatment.

Newly opened sterile masks were used for inhalation therapy in each child. In order to standardize the treatment, the 'Omron® CompAIR Pro NE-C900 Compressor Nebulizer' was used as a nebulizer. After each child, the infected materials of the VR glasses were removed with a surface disinfectant containing didecyldimethylammonium chloride and left in a disinfectant containing non-abrasive quarter ammonium carbonate, non-ionic surface active material and enzymatic complex, then rinsed with distilled water and waited until dry.

ELIGIBILITY:
Inclusion Criteria:

* Between 2-5 years old
* Children who need inhaler treatment (salbutamol)
* Children whose families give consent to participants the study

Exclusion Criteria:

* Children with neuromotor retardation,
* Visual and auditory problems,
* Underlying chronic diseases (bronchiolitis, chronic lung diseases other than asthma, congenital heart diseases, neurological diseases such as epilepsy),
* Obesity or malnutrition (to equalize the effectiveness of the drug dose),
* Adrenaline, budesonide or those who receive ipratropium bromide treatment,
* Those who will receive inhaler inhaler treatment for the first time,
* Those who have received inhaler treatment in the last 72 hours,
* Those who have a previous operation or sedative history,
* Those who have a fever above 37.5°C,
* Those who have used VR before,
* Patients with a saturation value below 92% at the time of admission,
* Those presenting with severe asthma attack,
* Those with respiratory failure symptoms,
* Patients with a score of 5 and above according to the bronchiolitis severity score
* Those under 2 years of age to avoid screen exposure patients (infants) and patients over 5 years old (school period)

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change in the FLACC (Face, Legs, Activity, Cry and Consolability ) pain scoring system | Baseline
  Changing pain scores by helping with uncomfortable procedures for children. The researchers used the FLACC (Face, Legs, Activity, Cry and Consolability ) scoring and scored between 0 and 10. A higher score indicated more pain and restlessness.

CONTACTS AND LOCATIONS:
Overall Officials: Berker Okay, M.D., Principal Investigator — Member
Locations (1):
- UHS Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD are available from the principal investigator upon reasonable request

REFERENCES:
- [Result] Das DA, Grimmer KA, Sparnon AL, McRae SE, Thomas BH. The efficacy of playing a virtual reality game in modulating pain for children with acute burn injuries: a randomized controlled trial [ISRCTN87413556]. BMC Pediatr. 2005 Mar 3;5(1):1. doi: 10.1186/1471-2431-5-1. PMID 15745448
- [Result] Mott J, Bucolo S, Cuttle L, Mill J, Hilder M, Miller K, Kimble RM. The efficacy of an augmented virtual reality system to alleviate pain in children undergoing burns dressing changes: a randomised controlled trial. Burns. 2008 Sep;34(6):803-8. doi: 10.1016/j.burns.2007.10.010. Epub 2008 Mar 5. PMID 18325675
- [Result] Ozalp Gerceker G, Ayar D, Ozdemir EZ, Bektas M. Effects of virtual reality on pain, fear and anxiety during blood draw in children aged 5-12 years old: A randomised controlled study. J Clin Nurs. 2020 Apr;29(7-8):1151-1161. doi: 10.1111/jocn.15173. Epub 2020 Jan 22. PMID 31889358
- [Result] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Result] Althumairi A, Sahwan M, Alsaleh S, Alabduljobar Z, Aljabri D. Virtual Reality: Is It Helping Children Cope with Fear and Pain During Vaccination? J Multidiscip Healthc. 2021 Sep 21;14:2625-2632. doi: 10.2147/JMDH.S327349. eCollection 2021. PMID 34584419